CLINICAL TRIAL: NCT02182206
Title: A Phase I Open Label Dose Escalation Study of Continuous Once-daily or Twice Daily Oral Treatment With BIBF 1120 in Patients With Advanced Solid Tumours
Brief Title: An Dose Escalation Study of Treatment With BIBF 1120 in Patients With Advanced Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1199.3
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Tumors
MeSH Terms: conditions — Neoplasms | interventions — nintedanib

ARMS (1):
- BIBF 1120 (Experimental)
  Interventions: Drug: BIBF 1120

INTERVENTIONS:
Drug: BIBF 1120

SUMMARY:
Maximum Tolerated Dose (MTD), safety, pharmacokinetics, efficacy of BIBF 1120, pharmacodynamic parameters (Dynamic Contrast-Enhanced Magnetic Resonance Imaging (DCE-MRI))

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with confirmed diagnosis of advanced, non resectable and/or metastatic solid tumours, who have failed conventional treatment, or for whom no therapy of proven efficacy exists, or who were not amenable to established forms of treatment
* Measurable tumour deposits by one or more techniques (X-ray), Computed Tomography (CT), Magnetic Resonance Imaging (MRI))
* At least one tumour lesion considered suitable for DCE-MRI as determined by discussion with centre radiologist. This lesion must not have been previously irradiated
* Age 18 years or older
* Life expectancy of at least three months
* Written informed consent given consistent with International Conference on Harmonisation-Good Clinical Practice (ICH-GCP) guidelines
* Eastern Cooperative Oncology Group (ECOG) performance score 0 or 1
* Patients completely recovered from any therapy-related toxicities from previous chemo-, hormone-, immuno-, or radiotherapies

Exclusion Criteria:

* Surgical procedures within four weeks of initiating treatment with the study drug, active ulcers, or injuries with incomplete wound healing
* Active infectious disease
* Uncontrolled, severe hypertension (diastolic BP (Blood Pressure) >100 mmHg, Systolic BP>180 mmHg)
* Gastrointestinal disorders that might have interfered with the resorption of the study drug
* Serious illness or concomitant non-oncological disease considered by the investigator to have been incompatible with the protocol
* Brain metastases requiring therapy
* Absolute neutrophil count less than 1500/mm3
* Platelet count less than 100 000/mm3
* Bilirubin greater than 1.5 mg/dl (>26 μmol/L, System International (SI) unit equivalent)
* Aspartate amino transferase (AST) and / or alanine amino transferase (ALT) greater than three times the upper limit of normal (if related to liver metastases greater than five times the upper limit of normal)
* Serum creatinine greater than 1.5 mg/dl (>132μmol/L, SI unit equivalent)
* Women and men who were sexually active and unwilling to use a medically acceptable method of contraception
* Pregnancy or breastfeeding
* Treatment with other investigational drugs; chemotherapy or hormone therapy (excluding Lutenizing Hormone Releasing Hormone (LHRH) agonists or bisphosphonates provided the lesion for MR (magnetic resonance) imaging did not arise from bone) or participation in another clinical study within the past four weeks before start of therapy or concomitantly with this study
* Patients unable to comply with the protocol
* Active alcohol or drug abuse
* History of autoimmune disease
* History of allergy to gadolinium or other intravenous (IV) contrast agent, indwelling medical devices or any other condition that would preclude MR scanning
* Patients requiring the ongoing use of dexamethasone, anti-histamines, anti-hypertensives or medications for the control of cardiac failure such as diuretics, where there was likely to be a need for alteration of dose during the study period. Dose adjustment of such medications may have independently altered vascular permeability or blood flow

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2003-06; Primary Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of BIBF 1120 | Up to 7 months
Incidence and intensity of Adverse Events according to common toxicity criteria (CTC) associated with increasing doses of BIBF 1120 | Up to 7 months

SECONDARY OUTCOMES:
Transfer constant (Ktrans) | Screening, day 2, 28 and 56
Extravascular-extracellular leakage volume (ve) | Screening, day 2, 28 and 56
Area under the gadolinium concentration time curve [0-60 seconds] (AUC[Gd]) | Screening, day 2, 28 and 56
Relative blood volume (rBV) | Screening, day 2, 28 and 56
Mean transit time (MTT) | Screening, day 2, 28 and 56
Relative blood flow (rBF) | Screening, day 2, 28 and 56
Volume of tumour showing contrast uptake | Screening, day 2, 28 and 56
Volume of tumour showing no contrast uptake | Screening, day 2, 28 and 56
Restricted diffusion | Screening, day 2, 28 and 56
Vessel size index | Screening, day 2, 28 and 56
Change in Eastern Cooperative Oncology Group (ECOG) performance score | Baseline, up to 7 months
Objective tumour responses according to the response evaluation criteria in solid tumour (RECIST) | Baseline, up to 7 months
Area under the plasma concentration-time curve following the first dose of uniform intervals τ over the time interval from zero to 24 hours (AUCτ,1) | up to 24 hours after the first dose on day 1
Area under the plasma concentration-time curve over the time interval from zero to the time of the last quantifiable drug concentration (AUC0-tz) | up to 24 hours after the first dose on day 1
Area under the plasma concentration-time curve over the time interval from zero extrapolated to infinity (AUC0-∞) | up to 24 hours after the first dose on day 1
Maximum measured plasma concentration following the first dose of uniform intervals τ (Cmax,1) | up to 24 hours after the first dose on day 1
Time from dosing to the maximum plasma concentration following the first dose of uniform intervals τ (tmax,1) | up to 24 hours after the first dose on day 1
Terminal half-life (t1/2) | up to 24 hours after the first dose on day 1
Mean residence time (MRTpo) | up to 24 hours after the first dose on day 1
Apparent clearance (CL/F) | up to 24 hours after the first dose on day 1
Apparent volume of distribution during the terminal phase (Vz/F) | up to 24 hours after the first dose on day 1
Area under the plasma concentration-time curve over the dosing interval τ (24 h) at steady state (AUCτ,ss) | up to 24 hours after drug administration on day 27
Predose plasma concentration at steady state immediately before dosing (Cpre,ss) | up to 24 hours after drug administration on day 27
Maximum plasma concentration at steady state over the dosing interval τ (Cmax,ss) | up to 24 hours after drug administration on day 27
Time from dosing to the maximum plasma concentration at steady state over the dosing interval τ (tmax,ss) | up to 24 hours after drug administration on day 27
Terminal half-life at steady state (t1/2,ss) | up to 24 hours after drug administration on day 27
Apparent clearance at steady state (CL/F,ss) | up to 24 hours after drug administration on day 27
Mean residence time at steady state (MRTpo,ss), | up to 24 hours after drug administration on day 27
Apparent volume of distribution during the terminal phase at steady state (Vz/F,ss) | up to 24 hours after drug administration on day 27
Accumulation ratio (RA) | up to 24 hours after drug administration on day 27
Minimum measured plasma concentration following the first dose of uniform intervals τ (Cmin,1) | up to 24 hours after the first dose on day 1
Time from first dosing to the minimum plasma concentration over the dosing interval τ (tmin,1) | up to 24 hours after the first dose on day 1
Minimum measured plasma concentration at steady state over the dosing interval τ (Cmin,ss) | up to 24 hours after drug administration on day 27
Time from last dosing to the minimum plasma concentration at steady state over the dosing interval τ (tmin,ss) | up to 24 hours after drug administration on day 27
Predose concentration of the 15th dose over the dosing interval τ (Cpre,15) | pre-dose on day 15

REFERENCES:
- [Derived] Lee CP, Taylor NJ, Attard G, Pacey S, Nathan PD, de Bono JS, Temple G, Bell S, Stefanic M, Stopfer P, Tang A, Koh DM, Collins DJ, d'Arcy J, Padhani AR, Leach MO, Judson IR, Rustin GJ. Phase I study of nintedanib incorporating dynamic contrast-enhanced magnetic resonance imaging in patients with advanced solid tumors. Oncologist. 2015 Apr;20(4):368-9. doi: 10.1634/theoncologist.2014-0250. Epub 2015 Mar 20. PMID 25795637